CLINICAL TRIAL: NCT05678491
Title: Endoscopic Treatment of Gastroesophageal Reflux Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 490996/2022
Record Dates: First submitted 2023-01-02; First posted 2023-01-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gastro Esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Patients with GERD will be examined at baseline and after three and six months. Variables of GERD will be compared between the three different time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic mucosal band ligation (Experimental): All 12 patients with GERD will undergo the same procedure. Multiple rubber bands will be used to ligate mucosa in the gastroesophageal junction and cardia in 3/4 of the circumference.
  Interventions: Other: Endoscopic mucosal band ligation

INTERVENTIONS:
Other: Endoscopic mucosal band ligation — The mucosa in 3/4 of the circumference of the gastroesophageal junction and cardia will be treated with mucosal band ligation left in place. This will be done during upper endoscopy in sedation. It is the endoscopic procedure that is being investigated.

SUMMARY:
Gastroesophageal reflux disease (GERD) occurs when stomach acid repeatedly flows back into the tube connecting your mouth and stomach (esophagus). This backwash (acid reflux) can irritate the inner lining of the esophagus. This is a particular problem after surgery to reduce obesity called gastric sleeve resection.

The goal of this small clinical trial is to examine the effect of endoscopic treatment of GERD by mucosal band ligation. The main questions it aims to answer are:

* Does the treatment affect gastroesophageal reflux assessed by measuring gastroesophageal reflux
* Does the treatment affect gastroesophageal reflux symptoms and ability to stop treatment with medication commonly used (proton pump inhibitors)

Participants (n=12) will be asked to undergo 24 h reflux examination and report symptoms of GERD. Suitable patients will be offered endoscopic treatment with band ligation of the inner lining of the lower esophagus and upper part of the stomach. The effects will be assessed three and six months after the procedure.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is very common after gastric sleeve resection and many patients are dependent on daily use of proton pump inhibitors (PPIs). The goal of this small clinical trial is to examine the effect of endoscopic treatment of GERD by mucosal band ligation.

Patients (n=12) with GERD satisfying inclusion and exclusion criteria will be invited to participate and the degree of gastroesophageal reflux will be assessed before treatment, and three and six months after the procedure. The results of the trial will be used to plan a larger study.

ELIGIBILITY:
Inclusion Criteria (all criteria must be fulfilled):

* Previous gastric sleeve resection
* GERD. GERD must be diagnosed by either endoscopic esophagitis or esophageal pH measurement with DeMeester score > 14.72 and pH <4 more than 4% of a 24-h period and symptom association probability (SAP) > 95%
* Subjective insufficient symptom control with PPI therapy once daily or intolerance to PPI or desire to stop PPI treatment and therefore willingness to undergo endoscopic treatment.

Exclusion Criteria:

* Hiatal hernia > 5 cm
* Age < 18_years
* Preexisting esophageal stricture
* Gastric stricture < 2 cm in diameter
* Anti-coagulant medication
* Use of platelet inhibitors other than acetylsalicylic acid
* Manometric indication of motility disorder
* Connective tissue diseases
* BMI > 35
* Liver cirrhosis
* Coronary heart disease
* Chronic obstructive pulmonary disease
* Other significant comorbidity
* Indication for long-term PPI use other than GERD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline esophageal 24 hour pH/impedance at 3 months | 3 months
  Esophageal pH/impedance will be measured by a catheter left in place for 24 hours
Change from baseline esophageal 24 hour pH/impedance at 6 months | 6 months
  Esophageal pH/impedance will be measured by a catheter left in place for 24 hours
Change from baseline symptoms of gastroesophageal reflux at 3 months | 3 months
  GERD Q score. Gastroesophageal reflux disease Questionnaire with minimum value 0 (no symptoms) and maximum value 18 (severe symptoms)
Change from baseline symptoms of gastroesophageal reflux at 6 months | 6 months
  GERD Q score. Gastroesophageal reflux disease Questionnaire with minimum value 0 (no symptoms) and maximum value 18 (severe symptoms)
Change from baseline in use of proton pump inhibitors (PPI) at 3 months | 3 months
  PPI use (number of days PPI was used during the period 7-14 days before the 3 months visit)
Change from baseline in use of proton pump inhibitors (PPI) at 6 months | 6 months
  PPI use (number of days PPI was used during the period 7-14 days before the 6 months visit)
Adverse events during the study period of 6 months | 6 months
  Adverse events or complications of the treatment will be registered during the study period

SECONDARY OUTCOMES:
Change from baseline in dysphagia at 3 months | 3 months
  Dysphagia assessed by Marks score. The minimum value is 0 (no dysphagia) and the maximum value is 6 (can not eat, which is the most severe symptom).
Change from baseline in dysphagia at 6 months | 6 months
  Dysphagia assessed by Marks score. The minimum value is 0 (no dysphagia) and the maximum value is 6 (can not eat, which is the most severe symptom).
Change from baseline in Hills flap valve at 3 months | 3 months
  The Hills flap valve assessed during endoscopy. Minimum value is 1 (good function) and the maximum value is 4 (poor function)
Change from baseline in Hills flap valve at 6 months | 6 months
  The Hills flap valve assessed during endoscopy. Minimum value is 1 (good function) and the maximum value is 4 (poor function)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Qvigstad, MD, PhD, Study Director — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
The plan is to publish all relevant data from this small trial with the detail level permitted by the local approval. Further data sharing will not be planned for.